CLINICAL TRIAL: NCT07351175
Title: Investigating The Potential Of A Hay-Aged Cheese To Reduce Cholesterol As Mediated By Changes In The Gut Microbiome: A Randomised Control Trial
Brief Title: Investigating The Potential Of A Hay-Aged Cheese To Reduce Cholesterol As Mediated By Changes In The Gut Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anisha Wijeyesekera (Other)
Responsible Party: Sponsor-Investigator, Anisha Wijeyesekera, Associate Professor, University of Reading
Organization: University of Reading (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UREC 25/39
Record Dates: First submitted 2026-01-02; First posted 2026-01-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cholesterol, Elevated
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be told which cheese they have been allocated, but the appearance of the cheese (hay-aged vs cheddar) will likely make it obvious to the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hay-aged cheese (Experimental): An artisan cheese aged in hay - this is a semi-hard cheese, aged for 9 months, with hay present on the rind.
  Interventions: Dietary Supplement: Hay-aged cheese
- Cheddar (Active Comparator): Industrial made cheddar, vintage aged. Vacuum packed.
  Interventions: Dietary Supplement: Cheddar control

INTERVENTIONS:
Dietary Supplement: Hay-aged cheese — This cheese is speculated to have both probiotic properties, from the starter cultures present in the cheese, and prebiotic properties, from the hay on the rind, making this cheese synbiotic.
  Arms: Hay-aged cheese
Dietary Supplement: Cheddar control — This cheese is an industrial made cheddar, it still has potential probiotic properties due to the starter cultures used, but no prebiotic potential.
  Arms: Cheddar

SUMMARY:
The goal of this intervention trial is to investigate the potential of an artisan cheese aged in hay to induce changes in the gut microbiota in a manner which mediates a reduction in total cholesterol in participants with elevated total cholesterol. The main questions it aims to answer are:

Does daily consumption of a hay aged cheese over 12 weeks reduce total cholesterol by at least 0.5mmol/l when compared the control cheese (cheddar)? Are changes in total cholesterol level reflected in changes in gut microbiota composition and activity as measured by deoxyribonucleic acid (DNA) sequencing of stool composition and short chain fatty acid levels in urine?

Participants will be asked to consume 30g portions of cheese every day for 12 weeks. This study is conducted in parallel, with participants either allocated onto the control arm (cheddar) or intervention arm (hay-aged cheese). Blood, stool, and urine samples will be taken throughout the trial, body mass index (BMI) and blood pressure will also be measured.

DETAILED DESCRIPTION:
Cheese production involves the use of starter culture bacteria, many of which are species with recognised probiotic potential. Additionally, the food matrix of protein and fat is thought to protect these cultures during human digestion, allowing them to reach the large intestine alive. Previous studies have indicated that cultures present in cheese can persist in the gut microbiome and exert a positive effect. Further studies have indicated that regular cheese consumption, despite having a high proportion of saturated fats, has been associated with lower cholesterol levels. This is thought to be mediated by the food matrix which reduces the release of fat during digestion, and recent work by the investigators has suggested that changes in the gut microbiota activity induced by cheese consumption may also have a role. This laboratory work has shown that cheese can boost the production of propionate (a microbially derived metabolite) in a gut model system, particularly a variety of cheese that is aged in hay (Witheridge-in-hay). Propionate in the gut is known to have a role in cholesterol regulation. The hypothesis is that cheese is a source of probiotics, and the hay on the rind of Witheridge-in-hay acts in a prebiotic manner; therefore this cheese is synbiotic and has the potential to confer multiple health benefits including reduced total cholesterol concentration mediated by a change in gut microbiota composition. In the proposed study, participants (ages 18-65, with elevated cholesterol between 5.5-7.5mmol/l) will consume a thirty-gram portion of cheese a day, either Witheridge-in-hay or cheddar as a control, for twelve weeks. Effects will be determined by collecting stool samples, urine, and blood from participants to measure bacterial composition, fermentation end products, and cholesterol levels respectively, as well as body mass index (BMI) measurements and blood pressure for further assessment of cardiovascular and weight gain effects. Samples will be collected at baseline, mid-intervention, and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 65 years old
* Regular consumer of cheese
* In generally good health but with total cholesterol level between 5.5-7.5 mmol/l and body mass index (BMI) between 18-32 kg/m2 at screening visit
* Willing and able to comply with study instructions

Exclusion Criteria:

* Use of antibiotics in the last 6 months prior to the study.
* Use of prebiotics, probiotics, laxatives, anti-spasmodic, anti-diarrhoeals, herb supplements in the last 4 weeks prior to or during the study period.
* Any chronic gut disorders/disease such as irritable bowel syndrome, inflammatory bowel disease, etc or other conditions that might affect the gut environment e.g. coeliac disease.
* High blood pressure, anaemia, high blood lipids (total cholesterol >7.5mmol/l), or inflammatory conditions
* Taking medication for anaemia, high blood pressure, high blood lipids , inflammatory conditions or depression
* Anyone diagnosed with vitamin deficiencies, diabetes, heart disease (previous stroke or heart attack) or have a pacemaker, kidney, bowel or liver diseases, cancer or hormone abnormalities.
* Pregnant, lactating, breast feeding or planning a pregnancy within the next 6 months
* Peri- or postmenopausal women
* Lost more than 3kg of body weight in the last 6 months
* Food allergies and intolerances
* Participants currently involved or will be involved in another clinical or food study in the previous 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in total cholesterol concentration | 12 weeks
  Total cholesterol levels will be measured at the beginning and end of the trial. Does the daily consumption of cheese have an effect on total cholesterol levels, and does consumption of a hay-aged cheese influence total cholesterol beyond that for cheddar?

SECONDARY OUTCOMES:
Change in faecal microbiota composition | 12 weeks
  Stool samples will be collected on 3 occasions throughout the trial. 16S sequencing will be used to assess changes in microbial populations in response to daily cheese consumption, comparing cheddar and the hay-aged cheese.
Change in production of SCFA by the gut microbiota | 12 weeks
  Gas chromatography will be used to analyse changes in SCFA content in stool and urine, collected on 3 and 5 occasions throughout the trial, respectively. This will help to assess the activity of the gut microbiota induced by the cheese intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anisha Wijeyesekera, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Department of Food and Nutritional Sciences, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No